CLINICAL TRIAL: NCT01590992
Title: Psychotherapy and Psychobiology of Somatoform Disorders (Globus Sensations): A Randomized Controlled Trial
Brief Title: Treatment of Globus Sensations With Psychotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other); Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT1_135328_A
Record Dates: First submitted 2012-04-11; First posted 2012-05-03 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Somatoform Disorders; Globus Hystericus
Keywords: Somatoform disorder; Functional Somatic Syndrome; Functional Somatic Symptoms; Somatic Symptom Disorder; globus sensation; globus pharynges; globus hystericus
MeSH Terms: conditions — Somatoform Disorders; Globus Sensation | interventions — Behavior Therapy; Implosive Therapy; Relaxation Therapy; Autogenic Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposure-based Psychotherapy for Somatic Symptoms (Experimental): First: 1-2 months waiting period; followed by: exposure-based psychotherapy
  Interventions: Behavioral: Exposure-based psychotherapy for somatic symptoms
- Relaxation Therapy (Active Comparator): First: 1-2 months waiting period; followed by: relaxation therapy
  Interventions: Behavioral: Relaxation therapy

INTERVENTIONS:
Behavioral: Exposure-based psychotherapy for somatic symptoms — Application of different types of exposure-based psychotherapeutic interventions (behavioral therapy), adapted for subjects with somatic symptoms (Somatoform Disorders/Functional Somatic Syndromes)
  Other Names: Behavioral therapy for somatic symptoms; Behavioural therapy for somatic symptoms; Exposure-therapy for somatic symptoms; Exposure-based psychotherapy for somatoform disorders; Behavioral therapy for somatoform disorders; Behavioural therapy for somatoform disorders; Exposure-therapy for somatoform disorders; Exposure-based psychotherapy for somatic symptom disorders; Behavioral therapy for somatic symptom disorders; Behavioural therapy for somatic symptom disorders; Exposure-therapy for somatic symptom disorders
  Arms: Exposure-based Psychotherapy for Somatic Symptoms
Behavioral: Relaxation therapy — Progressive muscle relaxation (Jacobson)
  Other Names: Progressive relaxation
  Arms: Relaxation Therapy

SUMMARY:
The purpose of this study is to determine whether psychotherapy (based on exposure techniques) is effective in the treatment of functional somatic symptoms (FSS)/Somatoform Disorders (as exemplified here in subjects with globus sensations in the throat).

DETAILED DESCRIPTION:
Functional somatic symptoms (FSS) and somatoform disorders are characterized by the presence of medically unexplained symptoms. They are among the most prevalent disorders in the general medical setting, leading to individual suffering and having huge impact on public health alike. Unfortunately, many patients still remain untreated and not all patients get better, even when receiving currently proposed treatments. The aim of the present project is twofold: First, we want to improve the understanding of risk factors and psychobiological processes leading to the development of FSS. Second, we will explore and evaluate new ways of treating subjects with FSS. Within the project, we will examine subjects with globus sensations in the throat, a very common und impairing form of FSS. The proposed study i) may provide insight into the development of FSS, thereby improving our way by which we recognize and diagnose subjects with FSS, and ii) may help fostering our understanding of how to better treat subjects suffering from FSS.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient spoken and written knowledge of German
* Presence of globus sensations and somatoform disorder
* Clinically significant impairment

Exclusion Criteria:

* Current (past 12 months) severe chronic physical illnesses, especially neurological, endocrine or metabolic diseases
* Current (past 12 months) substance dependence or eating disorder
* Lifetime history of psychotic disorder or bipolar disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2012-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression Scale - indirect (change from baseline) | Baseline, after waiting period (an expected average of 8 weeks after baseline), post-therapy (expected average of 16 weeks after baseline)
  German version
Glasgow-Edinburgh Throat Scale (change from baseline) | Baseline, after waiting period (exp. average of 8 weeks after baseline), post-therapy (exp. average of 16 weeks after baseline), Follow-up 1 (exp. average of 6 months after post-therapy), Follow-up 2 (exp. average of 24 months after post-therapy)
  German version
Functional Esophageal Disorder Module Interview (change from baseline) | Baseline, after waiting period (exp. average of 8 weeks after baseline), post-therapy (exp. average of 16 weeks after baseline), Follow-up 1 (exp. average of 6 months after post-therapy), Follow-up 2 (exp. average of 24 months after post-therapy)
  German version
Screening for somatoform disorder (SOMS-7) (change from baseline) | Baseline, after waiting period (exp. average of 8 weeks after baseline), post-therapy (exp. average of 16 weeks after baseline), Follow-up 1 (exp. average of 6 months after post-therapy), Follow-up 2 (exp. average of 24 months after post-therapy)

SECONDARY OUTCOMES:
Acceptance & Action Questionnaire (AAQ-II) | Baseline, after waiting period (exp. average of 8 weeks after baseline), post-therapy (exp. average of 16 weeks after baseline), Follow-up 1 (exp. average of 6 months after post-therapy), Follow-up 2 (exp. average of 24 months after post-therapy)
  German version
Fragebogen zu Körper und Gesundheit (FKG-SSAS) | Baseline, after waiting period (exp. average of 8 weeks after baseline), post-therapy (exp. average of 16 weeks after baseline), Follow-up 1 (exp. average of 6 months after post-therapy), Follow-up 2 (exp. average of 24 months after post-therapy)
Daily Symptom Exposure Interview | Baseline, after waiting period (exp. average of 8 weeks after baseline), post-therapy (exp. average of 16 weeks after baseline), Follow-up 1 (exp. average of 6 months after post-therapy), Follow-up 2 (exp. average of 24 months after post-therapy)
  German version
Hospital Anxiety and Depression Scale | Baseline, after waiting period (exp. average of 8 weeks after baseline), post-therapy (exp. average of 16 weeks after baseline), Follow-up 1 (exp. average of 6 months after post-therapy), Follow-up 2 (exp. average of 24 months after post-therapy)
  German version
Positive and Negative Affect Scale | Baseline, after waiting period (exp. average of 8 weeks after baseline), post-therapy (exp. average of 16 weeks after baseline), Follow-up 1 (exp. average of 6 months after post-therapy), Follow-up 2 (exp. average of 24 months after post-therapy)
Sheehan Disability Scale | Baseline, after waiting period (exp. average of 8 weeks after baseline), post-therapy (exp. average of 16 weeks after baseline), Follow-up 1 (exp. average of 6 months after post-therapy), Follow-up 2 (exp. average of 24 months after post-therapy)
  German version
Whiteley Index | Baseline, after waiting period (exp. average of 8 weeks after baseline), post-therapy (exp. average of 16 weeks after baseline), Follow-up 1 (exp. average of 6 months after post-therapy), Follow-up 2 (exp. average of 24 months after post-therapy)
  German version
Salivary Cortisol Awakening Response | Baseline, after waiting period (exp. average of 8 weeks after baseline), post-therapy (exp. average of 16 weeks after baseline)
DNA-methylation | Baseline, after waiting period (exp. average of 8 weeks after baseline), post-therapy (exp. average of 16 weeks after baseline)
Questions on adverse/side effects | Baseline, after waiting period (exp. average of 8 weeks after baseline), post-therapy (exp. average of 16 weeks after baseline), Follow-up 1 (exp. average of 6 months after post-therapy), Follow-up 2 (exp. average of 24 months after post-therapy)
psychophysiological reaction after symptom-relevant stimulus exposure | Baseline, after waiting period (exp. average of 8 weeks after baseline), post-therapy (exp. average of 16 weeks after baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Gunther Meinlschmidt, Ph.D., Study Director — University of Basel, Ruhr-University Bochum; Roselind Lieb, Ph.D., Study Director — University of Basel
Locations (1):
- University of Basel, Basel, Switzerland

REFERENCES:
- [Derived] Imperiale MN, Lieb R, Meinlschmidt G. Treatment-associated network dynamics in patients with globus sensations: a proof-of-concept study. Sci Rep. 2023 Sep 20;13(1):15615. doi: 10.1038/s41598-023-42186-y. PMID 37730963